CLINICAL TRIAL: NCT05301751
Title: A Multicenter, Open-Labeled, Phase 2a Study Evaluating the Safety, Tolerability, and Efficacy of Intravitreal AG-73305 in Patients With Diabetic Macular Edema
Brief Title: A Single Ascending Dose Cohort Study of AG-73305 in DME Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allgenesis Biotherapeutics Inc. (Industry)
Collaborators: Lexitas Pharma Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P2-73305-001
Record Dates: First submitted 2022-03-20; First posted 2022-03-31 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Macular Edema
Keywords: Allegenesis; Diabetic Macular Edema; AG-73305

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): 0.5 mg AG-73305 solution, single injection.
  Interventions: Biological: AG-73305
- Cohort 2 (Experimental): 1 mg AG-73305 solution, single injection.
  Interventions: Biological: AG-73305
- Cohort 3 (Experimental): 2 mg AG-73305 solution, single injection.
  Interventions: Biological: AG-73305
- Cohort 4 (Experimental): 4 mg AG-73305 solution, single injection.
  Interventions: Biological: AG-73305

INTERVENTIONS:
Biological: AG-73305 — drug product solution

SUMMARY:
This is a multi-centered, open-labeled, single ascending-dose-cohort study to evaluate the safety and efficacy of 4 dose cohorts of AG-73305 administered by intravitreal injection in patients with diabetic macular edema (DME).

The objectives of this study were to evaluate the safety, tolerability, duration of effect, systemic pharmacokinetic and immunogenicity profiles of ascending doses of AG-73305 administered by intravitreal injection to patients with DME. Pharmacodynamic endpoints (e.g., best-corrected visual acuity [BCVA], spectral domain optical coherence tomography [SD-OCT], and optical coherence tomography angiography [OCT-A]) were evaluated over 6 months post-treatment. The maximum tolerated dose or the highest administered dose was evaluated for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older at the screening visit
2. Prior diagnosis of diabetes mellitus (Type 1 or Type 2) as defined by World Health Organization or American Diabetes Association
3. Presence of center-involving DME in the study eye with CST ≥ 325 μm
4. Visual acuity loss in the study eye attributed to DME with screening and baseline ETDRS BCVA letter score of 20 to 55 (20/400 to 20/80 Snellen equivalent) in the sentinel patients and 35 to 70 (20/200 to 20/40 Snellen equivalent) in the non-sentinel patients
5. Cohort 1: Previously treated with an anti-VEGF in the study eye; Cohorts 2, 3, and 4: Previously treated or treatment-naïve to the study eye

Exclusion Criteria:

1. Uncontrolled diabetes mellitus, defined as hemoglobin A1c > 12.0% at Screening
2. Uncontrolled hypertension with systolic blood pressure ≥ 180 mmHg and/or diastolic blood pressure ≥ 100 mmHg at Screening or Baseline
3. Chronic renal disease
4. Any active infection in either eye
5. Any anti-vascular endothelial growth factor (VEGF) treatment in the study eye within 6 to 8 weeks prior to Baseline
6. Use of Ozurdex (dexamethasone) within 6 months prior to Baseline or any use of Iluvien (fluocinolone acetonide) in the study eye
7. Uncontrolled intraocular pressure (IOP), defined as an IOP > 25 mmHg, despite anti-glaucoma medications in the study eye at the time of screening or controlled glaucoma that requires management with > 2 topical hypotensive medications
8. Any anti-integrin therapy (e.g., Xiidra) within 60 days before baseline in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-12-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Center of Macula and Retina Disease, Winter Haven, Florida
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Valley Retina Institute, McAllen, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened based on the inclusion/exclusion criteria at 6 clinical sites in the US between May 2022 to December 2023.
Groups:
- Cohort 1: A single intravitreal (IVT) dose of 0.5 mg AG-73305
  AG-73305: AG-73305 Ophthalmic Solution
- Cohort 2: A single IVT dose of 1 mg AG-73305
  AG-73305: AG-73305 Ophthalmic Solution
- Cohort 3: A single IVT dose of 2 mg AG-73305
  AG-73305: AG-73305 Ophthalmic Solution
- Cohort 4: A single IVT dose of 4 mg AG-73305
  AG-73305: AG-73305 Ophthalmic Solution
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 3 | 6 | 8 | 8
Completed | 3 | 6 | 7 | 8
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 3 | 6 | 8 | 8 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 5 | 7 | 15
  >=65 years | 3 | 3 | 3 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (3.6) | 64.2 (9.9) | 59.6 (11.2) | 54.5 (14.7) | 60.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4 | 3 | 11
  Male | 3 | 2 | 4 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 4 | 3 | 9
  Not Hispanic or Latino | 2 | 5 | 4 | 5 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 3 | 6 | 8 | 7 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 8 | 8 | 25
Best-corrected Visual Acuity [Mean (Standard Deviation); unit: ETDRS letters] | 56.7 (1.5) | 48.7 (11.9) | 62.4 (5.4) | 63.0 (3.2) | 58.6 (8.8)
Central Subfield Thickness [Mean (Standard Deviation); unit: micrometers] | 522.017 (197.845) | 657.732 (169.990) | 444.818 (163.635) | 464.488 (140.934) | 511.475 (174.539)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA)
Description: BCVA assessments were performed at all visits utilizing ETDRS charts to assess changes in vision over time. The charts were designed for use at 4 meters. BCVA assessments were performed by certified technicians to minimize bias.
Time Frame: 1 month after dosing
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 6 | 8 | 8
ETDRS letters | 3.7 (1.2) | 9.2 (5.3) | 4.3 (3.9) | 7.7 (7.7)

2. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness (CST)
Description: SD-OCT imaging was performed at all visits utilizing Heidelberg Spectralis imaging equipment to assess changes over time in the structural details of the posterior segment of the eye. All images were graded by a central reading center.
Time Frame: 1 month after dosing
Measure: Mean (Standard Deviation); unit: μm
Units Other Than Participants: eyes
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 6 | 8 | 8
Number analyzed (eyes) | 3 | 6 | 8 | 8
μm | 2.287 (9.819) | -263.167 (221.986) | -70.443 (175.147) | -50.571 (108.694)

ADVERSE EVENTS:
Time Frame: 6 months (24 weeks)
Groups:
- Cohort 1: A single intravitreal (IVT) dose of 0.5 mg AG-73305
- Cohort 2: A single IVT dose of 1 mg AG-73305
- Cohort 3: A single IVT dose of 2 mg AG-73305
- Cohort 4: A single IVT dose of 4 mg AG-73305
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 1/8 | 1/8
Other Adverse Events (participants affected / at risk) | 3/3 | 4/6 | 6/8 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=6) | Cohort 3 (N=8) | Cohort 4 (N=8)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The Investigator reported that the event was severe in intensity, and was unrelated to AG-73305.
Kidney failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) — The Investigator reported that the event was severe in intensity, and was unrelated to AG-73305.
Acute respiratory failure with hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) — The Investigator reported that the event was severe in intensity, and was unrelated to AG-73305.
Congestive heart failure excerbation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — The Investigator reported that the event was severe in intensity, and was unrelated to AG-73305.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=6) | Cohort 3 (N=8) | Cohort 4 (N=8)
Iridocyclitis (drug related) (Eye disorders) | 2 (2) | 4 (4) | 3 (4) | 4 (6)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) — The Investigator reported that the event was not related to AG-73305.
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) — The Investigator reported that the event was not related to AG-73305.
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — The Investigator reported that the event was not related to AG-73305.
anterior chamber inflammation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The Investigator reported that the event was not related to AG-73305.
Iridocylitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) — The Investigator reported that the event was not related to AG-73305.

LIMITATIONS AND CAVEATS:
Study was designed to assess safety, and efficacy endpoints were not statistically powered. Results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT05301751/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT05301751/SAP_001.pdf